CLINICAL TRIAL: NCT03314649
Title: Prospective Observational Study of Peritoneal Lavage for Early Detecting Gene Mutation of Peritoneal Metastasis of Gastric Cancer
Brief Title: Peritoneal Lavage for Early Detecting Gene Mutation of Peritoneal Metastasis of Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Dazhi Xu, Professor, Fudan University
Other Study IDs: CGCG003
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Gastric Cancer
Keywords: Peritoneal Lavage, Gene Mutation, Peritoneal Metastasis,Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor biopsy, peritoneal lavage
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational study: Patients with gastric cancer and non-cancerous disease planned to have laparotomy
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Lavage of the Peritoneal Cavity

SUMMARY:
Our study aims to improve sensitivity and accuracy of detecting abdominal free cancer cells in patients with gastric cancer.

DETAILED DESCRIPTION:
Gastric cancer (GC) remains one of the most common causes of cancer-related mortality worldwide. Surgery has always been considered as the most effective treatment for GC. Peritoneal metastasis is the common pattern of postoperative recurrence, especially patients with T4 stage or serosal invasion. What is worse, patients with peritoneal metastasis have a poor prognosis. However, it is often difficult to diagnose peritoneal metastasis at an early stage. As we know, the implantation of peritoneal free cancer cells exfoliating from serosa-invasive tumors is main reason of peritoneal seeding. Cytological examination of peritoneal lavage fluid is always performed to predict peritoneal micrometastases. However, more than half of patients with negative cytological results develop peritoneal recurrence. Low sensitivity and poor negative predictive value of this method have heralded the development of advanced techniques in detecting peritoneal free cancer cells.

In this study, novel genetic techniques will be used to detect mutated DNA of shed cancer cells in abdominal cavity. The present clinical trial aims to find a better tool to detect abdominal micrometastasis in GC patients, which may become a valid clinical index to predict postoperative relapse and direct treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Lower age limit of research subjects 18 years old and upper age limit of 80 years old.
2. PS (ECOG) of 0 or 1 and expected to survive more than 6 months.
3. Written informed consent from the patient.
4. Patients suffering gastric cancer and non-cancerous disease planned to have laparotomy.

Exclusion Criteria:

1. Female in pregnancy or lactation. 2. Patients participating in any other clinical trials currently，or participated in other trails within 1 months. 3. Patients with poor compliance or considered to be poor compliance.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering gastric cancer and non-cancerous disease planned to have laparotomy.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
prognostic molecular markers | 3-year
  prognostic molecular markers

SECONDARY OUTCOMES:
OS | 3-year
  Overall survival
DFS | 3-year
  Disease-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center of Sun Yat-sen University, Guangzhou, Guangdong, China